CLINICAL TRIAL: NCT05313386
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-controlled, Ascending Starting Dose Finding, Safety, and Efficacy Study of BXCL501 in Agitation Associated With Delirium in ICU Patients.
Brief Title: Study of BXCL501 In Agitation Associated With Delirium in ICU Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped early, before enrolling its first participant
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXCL501-202
Record Dates: First submitted 2021-03-31; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Agitation; Delirium
MeSH Terms: conditions — Psychomotor Agitation; Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Cohorts will be enrolled sequentially in this dose escalating design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1- 120 Micrograms (Experimental): 120 Micrograms film or Placebo film are given to patients in 3:1 ratio respectively.
  Repeat doses may be administered in increments of 120 μg every 3 to 6 hours post first dose (StartD) only if the RASS score remains ≥ +1. For subjects 65 years and older, repeat doses may start in increments of 60 μg every 3 to 6 hours post first dose only if RASS is still ≥+1.
  Interventions: Drug: BXCL501; Drug: Placebo film
- Cohort 2- 180 Micrograms (Experimental): 180 Micrograms film or Placebo film are given to patients in 3:1 ratio respectively.
  Repeat doses may be administered in increments of 120 μg every 3 to 6 hours post first dose (StartD) only if the RASS score remains ≥ +1. For subjects 65 years and older, repeat doses may start in increments of 60 μg every 3 to 6 hours post first dose only if RASS is still ≥+1.
  Interventions: Drug: BXCL501; Drug: Placebo film
- Cohort 3- 240 Micrograms (Experimental): Two 120 Micrograms films or two Placebo films are given to patients in 3:1 ratio respectively.
  Repeat doses may be administered in increments of 120 μg every 3 to 6 hours post first dose (StartD) only if the RASS score remains ≥ +1. For subjects 65 years and older, repeat doses may start in increments of 60 μg every 3 to 6 hours post first dose only if RASS is still ≥+1.
  Interventions: Drug: BXCL501; Drug: Placebo film
- Cohort 4- 300 Micrograms (Experimental): One 120 Micrograms film and one 180 Micrograms film or two Placebo films are given to patients in 3:1 ratio respectively.
  Repeat doses may be administered in increments of 120 μg every 3 to 6 hours post first dose (StartD) only if the RASS score remains ≥ +1. For subjects 65 years and older, repeat doses may start in increments of 60 μg every 3 to 6 hours post first dose only if RASS is still ≥+1.
  Interventions: Drug: BXCL501; Drug: Placebo film

INTERVENTIONS:
Drug: BXCL501 — BXCL501 is given in a film form
  Other Names: Dexmedetomidine
Drug: Placebo film — Placebo is given in a film form

SUMMARY:
This study is designed to determine and evaluate the optimal BXCL501 starting dose (StartD) that will safely and effectively reduce agitation associated with delirium in ICU patients. This is an ascending adaptive dose study evaluating the safety and efficacy of four potential starting doses of BXCL501 (120 μg, 180 μg, 240 μg, and 300 μg) in reducing agitation levels in adult ICU patients with delirium. For subjects 65 years of age and older, the potential doses will be reduced 50% in line with the Precedex (reference drug) label. The purpose of this clinical trial is to identify an optimally safe and effective BXCL501

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, ascending starting dose finding study assessing safety, efficacy, tolerability and PK of BXCL501 in four starting dose cohort groups to reduce agitation levels associated with delirium in patients within the ICU setting. Evaluation of four BXCL501 starting doses compared to placebo will be conducted according to the following ascending doses: Cohort 1 (120 μg or placebo); Cohort 2 (180 μg or placebo); Cohort 3 (240 μg or placebo); Cohort 4 (300 μg or placebo). For subjects 65 years of age and older, the starting doses in each cohort will be reduced 50% in line with the Precedex (reference drug) label. Safety, efficacy, and tolerability will be assessed throughout the treatment period at various timepoints. Subjects will receive the first starting dose (BXCL501 or placebo) when Baseline RASS score is ≥ +1. Repeat doses may be administered in increments of 120 μg every 3 to 6 hours post first dose (StartD) only if the RASS score remains ≥ +1. For subjects 65 years and older, repeat doses may start in increments of 60 μg every 3 to 6 hours post first dose only if RASS is still ≥+1.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Enrollment (Informed Consent):

1. ICU admitted male and female patients, ≥ 18 years, COVID 19 (+) and (-)
2. Subject or legally appointed representative (LAR) able to read, understand and provide informed consent, or to provide assent

   Inclusion Criteria for Randomization:
3. Positive CAM-ICU
4. RASS score ≥ +1
5. Subject judged to be likely capable of self-administration

Exclusion Criteria:

1. Clinically significant ECG changes, brady- and tachyarrhythmias, QTc prolongation
2. Hepatic dysfunction
3. Pregnancy
4. Known allergy to Dexmedetomidine or Haloperidol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-02-21 (Estimated); Study Completion 2022-02-21 (Estimated)

PRIMARY OUTCOMES:
2-point or greater drop in RASS | 120 minutes
  Identification of the dose leading to a 2-point or greater drop in RASS at 2 hours after starting dose administration, with initial RASS not ≤ -3

SECONDARY OUTCOMES:
The time to which a 2-point drop is seen in RASS score after starting dose administration | 24 Hours
  The time to which a 2-point drop is seen in RASS score after starting dose administration.
Overall delirium improvement as measured by the CAM-ICU-7 Total Score during ICU stay | 24 Hours
  Overall delirium improvement as measured by the CAM-ICU-7 Total Score during ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- BioXcel Clinical Research Site, Nashville, Tennessee, United States